CLINICAL TRIAL: NCT05518500
Title: A Deep Longitudinal Analysis of Next Generation Influenza Vaccines in Older Adults
Acronym: FluVax3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Jackson Laboratory (Other)
Collaborators: UConn Health (Other); Icahn School of Medicine at Mount Sinai (Other); Weill Medical College of Cornell University (Other); University of Chicago (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Duygu Ucar, Ph.D., Associate Professor, The Jackson Laboratory
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-179J-1; U01AI165452 (NIH)
Record Dates: First submitted 2022-08-02; First posted 2022-08-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aging; Influenza Vaccine; Dendritic Cell; Vaccine Response
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Older Adults (Experimental): Will receive FDA-approved influenza vaccine (Fluzone HD Year 1, FLUAD Year 2, Flublok Quadrivalent Year 3)
  Interventions: Biological: Flu Vaccine (Year 1); Biological: Flu Vaccine (Year 2); Biological: Flu Vaccine (Year 3)

INTERVENTIONS:
Biological: Flu Vaccine (Year 1) — Participants will receive Fluzone® Quadrivalent High-Dose in the 2022-2023 flu season.
  Other Names: Fluzone® Quadrivalent High-Dose
Biological: Flu Vaccine (Year 2) — Participants will receive FLUAD® Quadrivalent in the 2023-2024 flu season.
  Other Names: FLUAD
Biological: Flu Vaccine (Year 3) — Participants will receive Flublok Quadrivalent in the 2024-2025 flu season.
  Other Names: Flublok Quadrivalent

SUMMARY:
This is a prospective, single-arm study designed to understand the mechanisms that lead to a loss of response to influenza vaccine in older adults. The investigators will recruit and longitudinally follow a cohort of 75 older adults (65 years and older) who will receive three different influenza vaccines over three annual influenza seasons. Blood samples will be collected from the participants at sixteen study visits over three years. Nasal swab and stool samples will also be collected from participants at seven time-points across the study period. The study is not designed to assess safety or tolerability of the influenza vaccines administered as part of this study.

DETAILED DESCRIPTION:
This prospective, single-arm study is designed to understand the mechanisms that lead to a loss of response to influenza vaccine in older adults through the establishment of the FluVax3 cohort of healthy older adults. In this study, the investigators will perform comprehensive profiling of blood antibodies and immune cells over time, and associate specific age-related immune alterations with vaccine responder or non-responder status. This will allow the investigators to pinpoint biological pathways that can be targeted to enhance vaccine efficacy and that can also help the investigators progress towards developing a universal influenza vaccine. The results are expected to provide the foundation for new approaches to improve overall vaccine efficacy and protection in older adults, an outcome of significant public health relevance considering the vulnerability of this population.

In this study, up to seventy-five (75) healthy adults aged 65 years and older who have not received influenza vaccination for the approaching influenza season will be enrolled in the study and vaccinated with influenza vaccines approved by the U.S Food and Drug Administration (FDA) and recommended by the Centers for Disease Control and Prevention (CDC) for individuals ≥65 years. All participants receive influenza vaccine during the 2022-23, 2023-24, and 2024-25 influenza seasons. Participants will receive Fluzone® Quadrivalent High-Dose vaccine during the 2022-23 flu season, FLUAD® Quadrivalent during the 2023-24 flu season and Flublok Quadrivalent in the 2024-2025 flu season. The study sample will be drawn from the population of healthy older participants in the catchment area of UConn Health in Farmington, CT.

Study participation will involve six study visits around the flu vaccine each year and one final study visit for a total of nineteen study visits over three years. Blood samples will be collected at sixteen study visits for transcriptional, epigenetic and biological analyses pre- and post-vaccination. Nasal swab and stool samples will also be collected from participants at seven time-points across the study period. These microbiome samples will be stored and used in future research. The study is not designed to assess safety or tolerability of the influenza vaccines administered as part of this proposed study.

This project will yield an unparalleled dataset from healthy older adults that will be used to identify fundamental mechanisms, cell populations, and pathways associated with durable protective antibody immune responses, and lack thereof, upon influenza vaccination. In sum, this study will reveal the mechanistic alterations that explain the heterogeneity in response to vaccines observed in older individuals. Understanding this heterogeneity opens the possibility of stratifying older adults for personalized vaccines. In addition, understanding the mechanistic overlap between the correlates of responsiveness to three different influenza vaccines will advance the ultimate development of a universal influenza vaccine, which is a key focus of NIAID's influenza research program. Finally, this study will generate a considerable amount of transcriptional and functional data related to the outputs of key innate immune and T/B-cell subsets involved in responses to influenza vaccines in older adults. These data will collectively become an important resource for future studies focused on the older adult immune system in health and disease.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English
* Male or Female, 65 years and older by date of enrollment
* Weight of 110 lbs or greater
* Has received influenza vaccine in the past seasons without severe adverse reactions
* Willing to receive an FDA-approved age-appropriate and CDC-recommended influenza vaccine for each of the 2022-23, 2023-24, and 2024-25 influenza seasons
* Willing to withhold all other vaccinations 2 weeks prior and 2 weeks after flu vaccination for the 2022-23, 2023-24, and 2024-25 influenza seasons
* Willing and available to participate in 19 study visits over three years around influenza vaccination
* Willing to provide blood samples at sixteen visits over three years
* Willing to agree to genomic testing of samples and sharing of de-identified genomic data generated from samples at the conclusion of the research

Exclusion Criteria:

* Received any vaccine (shingles, pneumococcal, COVID, etc.) within 2 weeks of anticipated flu vaccination for the 2022-23, 2023-24, and 2024-25 influenza seasons.
* Has already received an influenza vaccine for the approaching influenza season (2022-23)
* Has known allergy to eggs or any component of the flu vaccine. [Although the Advisory Committee on Immunization Practices (ACIP) has concluded that a history of anaphylactic/anaphylactoid or severe allergic reaction to eggs should no longer be considered a contraindication to vaccination with any age-appropriate vaccine, for the purposes of this research study we elected to exclude individuals with these allergies]
* History of Guillain-Barre syndrome (GBS)
* Body temperature greater than 100.3°F (38°C) on date of vaccination or within 2 days prior to vaccination by participant report (study entry may be delayed to meet this requirement)
* Rockwood Frailty Index score of >0.21
* Known history of any of the following co-morbid conditions:

  * Chronic or recent (within past 2 months) infection requiring oral or intravenous antibiotics, antifungals, or antivirals
  * Cancer other than basal cell carcinoma requiring active surgical or medical treatment (chemotherapy or radiation therapy)
  * Congestive Heart Failure
  * Ischemic Heart Disease
  * Congenital abnormalities (PI to evaluate)
  * Paget's disease
  * Renal failure requiring ongoing dialysis
  * Chronic obstructive pulmonary disease, emphysema, or asthma
  * Severe autoimmune disease requiring biological therapy
  * Diabetes mellitus requiring insulin
  * Use of medicines during past 6 months known to alter immune response such as high-dose corticosteroids (≥ 10 mg/day of prednisone or equivalent)
  * HIV, AIDS or other immunodeficiency disorders
  * Recent (≤ 3 months) severe trauma or major surgery (PI to evaluate)
  * Current substance and/or alcohol abuse
* Patients currently residing in the Department of Correction
* Inability to comply with the protocol requirements
* Any other condition that, in the opinion of the PI, might interfere with study objectives

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Antibody Responses to Influenza Vaccine Year One | Baseline, Day 35, Day 180
  In year one, healthy older participants will receive Fluzone Quadrivalent HD vaccine. Longitudinal blood samples will be collected and influenza-specific antibody responses will be assessed. Change in antibody response will be measured using Hemagglutination Inhibition (HAI) from baseline to day 35 and day 180.
Change in Antibody Responses to Influenza Vaccine Year Two | Baseline, Day 35, Day 180
  In year two, healthy older participants will receive FLUAD vaccine. Longitudinal blood samples will be collected and influenza-specific antibody responses will be assessed. Change in antibody response will be measured using Hemagglutination Inhibition (HAI) from baseline to day 35 and day 180.
Change in Antibody Responses to Influenza Vaccine Year Three | Baseline, Day 35, Day 180
  In year three, healthy older participants will receive Flublok Quadrivalent. Longitudinal blood samples will be collected and influenza-specific antibody responses will be assessed. Change in antibody response will be measured using Hemagglutination Inhibition (HAI) from baseline to day 35 and day 180.

SECONDARY OUTCOMES:
Evaluate changes in functional status of immune cells in response to Influenza Vaccine in Year One | Baseline, Day 7, Day 35
  Evaluate changes in functional status of immune cells in older participants following administration of Fluzone Quadrivalent HD vaccine. A longitudinal analysis of different cell populations (B Cells, Functional T/B Cells, and monoclonal antibodies) in whole blood samples will be analyzed at baseline and 35 days post vaccination using single cell assays and ELISA.
Evaluate changes in functional status of immune cells in response to Influenza Vaccine in Year Two | Baseline, Day 7, Day 35
  Evaluate changes in functional status of immune cells in older participants following administration of FLUAD vaccine. A longitudinal analysis of different cell populations (B Cells, Functional T/B Cells, and monoclonal antibodies) in whole blood samples will be analyzed at baseline and 35 days post vaccination using single cell assays and ELISA.
Evaluate changes in functional status of immune cells in response to Influenza Vaccine in Year Three | Baseline, Day 7, Day 35
  Evaluate changes in functional status of immune cells in older participants following administration of Flublok Quadrivalent. A longitudinal analysis of different cell populations (B Cells, Functional T/B Cells, and monoclonal antibodies) in whole blood samples will be analyzed at baseline and 35 days post vaccination using single cell assays and ELISA.
Number of genes upregulated in response to Influenza Vaccine in Year One | Baseline, Day1, Day 7
  RNA-seq and scRNA-seq will be used to assess the number of genes upregulated in response to Fluzone Quadrivalent HD vaccination.
Number of genes upregulated in response to Influenza Vaccine in Year Two | Baseline, Day 1, Day 7
  RNA-seq and scRNA-seq will be used to assess the number of genes upregulated in response to FLUAD vaccination.
Number of genes upregulated in response to Influenza Vaccine in Year Three | Baseline, Day1, Day 7
  RNA-seq and scRNA-seq will be used to assess the number of genes upregulated in response to Flublok Quadrivalent.
Number of chromatin accessibility regions activated in response to Influenza Vaccine in Year One | Baseline, Day1, Day 7
  snATAC-seq will be used to assess the number of open chromatin regions activated in response to Fluzone Quadrivalent HD vaccination.
Number of chromatin accessibility regions activated in response to Influenza Vaccine in Year Two | Baseline, Day1, Day 7
  snATAC-seq will be used to assess the number of open chromatin regions activated in response to FLUAD vaccination.
Number of chromatin accessibility regions activated in response to Influenza Vaccine in Year Three | Baseline, Day1, Day 7
  snATAC-seq will be used to assess the number of open chromatin regions activated in response to Flublok Quadrivalent influenza vaccination.
Changes in number of cDCs, Tfh, Th10, and B lymphocytes in response to Influenza Vaccine in Year One | Baseline, Day1, Day 7, Day 35, Day 180
  Flow cytometry will be used to assess cell compositional changes in PBMCs and immune cell subsets (cDCs, Tfh, Th10, and B lymphocytes) in response to Fluzone Quadrivalent HD vaccination.
Changes in number of cDCs, Tfh, Th10, and B lymphocytes in response to Influenza Vaccine in Year Two | Baseline, Day1, Day 7, Day 35, Day 180
  Flow cytometry will be used to assess cell compositional changes in PBMCs and immune cell subsets (cDCs, Tfh, Th10, and B lymphocytes) in response to FLUAD vaccination.
Changes in number of cDCs, Tfh, Th10, and B lymphocytes in response to Influenza Vaccine in Year Three | Baseline, Day1, Day 7, Day 35, Day 180
  Flow cytometry will be used to assess cell compositional changes in PBMCs and immune cell subsets (cDCs, Tfh, Th10, and B lymphocytes) in response to Flublok Quadrivalent influenza vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: George Kuchel, MD, FRCP, Principal Investigator — UConn Center on Aging
Locations (1):
- UConn Health, Center On Aging, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will provide permission within the ICF for sharing their randomly recoded (new code that is different than the study code) genomic data in controlled access scientific databases.
  Participants will provide permission within the ICF for sharing of randomly recoded (new code that is different than the study code) residual samples and linked data with other researchers to be used in future research studies.
Time Frame: Conclusion of the study
Access Criteria: Pending dbGaP/ImmPORT registration